CLINICAL TRIAL: NCT04878926
Title: IV Sedation Plus TAP Block for Placement of Percutaneous Endoscopic Gastrostomy Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DTH:18001
Record Dates: First submitted 2021-05-02; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2018-03

CONDITIONS: Transversus Abdominis Plane (TAP) Block
Keywords: Anesthesia; Endoscopic; Percutaneous gastrostomy; Sedation; TAP block
MeSH Terms: conditions — Bites and Stings | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (n=30) (Active Comparator): IV Sedation + TAP block
  Interventions: Procedure: IV midazolam and propofol-based sedation combined with ultrasound-guided, left side TAP block
- Group B (n=30) (Active Comparator): IV Sedation + LA infiltration
  Interventions: Procedure: IV midazolam and propofol-based sedation with Local Anesthetic infiltration

INTERVENTIONS:
Procedure: IV midazolam and propofol-based sedation combined with ultrasound-guided, left side TAP block — IV midazolam and propofol-based sedation combined with ultrasound-guided, left side TAP block
  Arms: Group A (n=30)
Procedure: IV midazolam and propofol-based sedation with Local Anesthetic infiltration — IV midazolam and propofol-based sedation with Local Anesthetic infiltration
  Arms: Group B (n=30)

SUMMARY:
Objective: To determine the effectiveness and safety of IV sedation combined with ultrasound-guided, left side transversus abdominis plane (TAP) block versus combination with local anesthetic (LA) infiltration for Percutaneous Endoscopic Gastrostomy (PEG) tube placement.

Background: The procedure used to be done with general anesthesia or IV sedation with LA infiltration, but the use of IV sedation with TAP block may be another option.

Patients and Methods: This was a prospective randomized study including 60 patients, requiring long-term nutritional support, underwent the PEG procedure at the GIT endoscopy unit at our Hospital. Patients were randomly allocated into two equal groups, in group A; procedures were performed with IV midazolam and propofol-based sedation combined with ultrasound-guided, left side TAP block, while in group B; procedures were performed with IV midazolam and propofol-based sedation with LA infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring long-term nutritional support
* American Society of Anesthesiologists (ASA) physical status II-III
* Age ≥ 6 years

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status > III
* Patients younger than 6 years
* Previous PEG placement
* Allergy to local anesthetics
* Patient refusal

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Successful completion of the operation | 20 minutes after introducing the endoscope in the patient mouth
  Successful placement of percutaneous endoscopic gastrostomy Tube

SECONDARY OUTCOMES:
Mean and Standard deviation of Heart Rate (beat/minute)(mean±SD) | 30 minutes after patients entered the endoscopy room
  After patients entered the endoscopy room (T0), 10 minutes after beginning of operation (T1), and at PACU (T2)
Mean and Standard deviation of Blood Pressure (mmHg)(mean±SD) | 30 minutes after patients entered the endoscopy room
  After patients entered the endoscopy room (T0), 10 minutes after beginning of operation (T1), and at PACU (T2)
Mean and Standard deviation of Oxygen Saturation (SpO2) (%)(mean±SD) | 30 minutes after patients entered the endoscopy room
  After patients entered the endoscopy room (T0), 10 minutes after beginning of operation (T1), and at PACU (T2)
Number of participants and Rate of Anesthesia-related Complications | 24 hours after the end of operation
  Number of participants and Rate of: Hypertension or Hypotension (increase or decrease in blood pressure by 20% from baseline); Tachycardia (Heart Rate > 100 beat/minute) or Bradycardia (Heart Rate < 60 beat/minute); Any cardiac arrhythmias; Hypoxemia (Oxygen desaturation, SpO2 < 90%), Failure of TAP block, Local Anesthetic toxicity, Intraperitoneal injection and Bowel injury
Median and Range of Numeric Pain Rating Scale (NPRS) | 24 hours after the end of operation
  NPRS measures the severity of pain, it is a 11 point scale from 0-10; where 0=No pain and 10=Worst possible pain (2 hours, and 24 hours after operation)
Mean and Standard deviation of Hospital stay duration (hour)(mean±SD) | 48 hours after entering the endoscopy unit
  Time interval from entering the hospital till discharge
Number of participants and Rate of Patients' Satisfaction of the service | 48 hours after entering the endoscopy unit
  YES/NO questionnaire for Patients' Satisfaction of the service

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt